CLINICAL TRIAL: NCT00019773
Title: Pilot Study of Oxaliplatin in Combination With Capecitabine in Adult Cancer Patients
Brief Title: Oxaliplatin Plus Capecitabine in Treating Patients With Colorectal, Appendix, or Small Bowel Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067201; NCI-99-C-0117; MB-NAVY-99-01; NCI-T99-0011; NCT00001817 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2003-04

CONDITIONS: Carcinoma of the Appendix; Colorectal Cancer; Small Intestine Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage 0 colon cancer; stage 0 rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; recurrent small intestine cancer; carcinoma of the appendix
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining oxaliplatin with capecitabine in treating patients who have colorectal, appendix, or small bowel cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of capecitabine when administered with oxaliplatin in patients with colorectal, appendiceal, or small bowel cancer.
* Determine the clinical toxic effects associated with this regimen in these patients.
* Characterize the molecular profile of tumor tissue obtained prior to study entry for determinants of sensitivity to this regimen in this patient population.
* Characterize the molecular profile of a surrogate normal tissue (bone marrow aspirate) obtained prior to treatment and assess any potential drug-associated induction of DNA damage and inhibition of thymidylate synthase with a repeat bone marrow aspirate during therapy.
* Assess any clinical activity of this regimen in this patient population.

OUTLINE: This is a dose-escalation study of capecitabine.

Patients receive oxaliplatin IV over 2 hours on day 1 followed by oral capecitabine twice daily on days 1-5 and 8-12. Courses repeat every 3 weeks in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 6 months.

PROJECTED ACCRUAL: A total of 106 patients will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal, appendiceal, or small bowel cancer
* Measurable disease
* No progression after prior capecitabine
* No brain metastases or leptomeningeal carcinomatosis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No sensory neuropathy
* No history of allergy to platinum compounds
* No history of allergy to antiemetics appropriate for administration during study
* No history of intolerance to fluorouracil
* No uncontrolled concurrent illness that would preclude study entry
* No ongoing or active infection requiring IV antibiotics
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* Recovered from prior chemotherapy
* No more than 2 prior systemic chemotherapy regimens for metastatic disease
* At least 6 weeks since prior nitrosoureas or mitomycin
* At least 8 weeks since prior eniluracil
* At least 3 months since prior suramin
* At least 4 weeks since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Recovered from prior radiotherapy
* At least 2 weeks since prior radiotherapy to no more than 20% of bone marrow reserve
* At least 4 weeks since prior radiotherapy to at least 21% of bone marrow reserve

Surgery:

* Recovered from prior surgery

Other:

* At least 4 weeks since prior sorivudine or brivudine and recovered
* No concurrent sorivudine or brivudine
* No other concurrent investigational agents
* No other concurrent anticancer therapy or commercial agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szabo, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Lehky TJ, Leonard GD, Wilson RH, Grem JL, Floeter MK. Oxaliplatin-induced neurotoxicity: acute hyperexcitability and chronic neuropathy. Muscle Nerve. 2004 Mar;29(3):387-92. doi: 10.1002/mus.10559. PMID 14981738
- [Result] Leonard G, Wright M, Quinn M, et al.: Survey of oxaliplatin-associated neurotoxicity with an interview-based questionnaire. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-3018, 2003.
- [Result] Wilson RH, Lehky T, Thomas RR, Quinn MG, Floeter MK, Grem JL. Acute oxaliplatin-induced peripheral nerve hyperexcitability. J Clin Oncol. 2002 Apr 1;20(7):1767-74. doi: 10.1200/JCO.2002.07.056. PMID 11919233
- [Result] Thomas R, Quinn M, Wilson R, et al.: A phase I trial of capecitabine (CAPE) & oxaliplatin (OHP). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-530, 2001.